CLINICAL TRIAL: NCT06968156
Title: The Effect of Monocyte Values Accompanied by Lymphopenia on the Prognosis of Patients Diagnosed With COVID-19
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Naime Yalçın, Anesthesiology and Reanimation specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KAEK/2021.04.142
Record Dates: First submitted 2025-05-01; First posted 2025-05-13 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: COVID 19; Lymphopenia Due to COVID-19; Monocyte
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group monocytopenia
- Group control
- Group monocytosis

SUMMARY:
Recent studies have shown that lymphopenia with cytokine storm syndrome is frequently found in COVID-19 patients. These features may suggest that the modified immune system plays a key role in determining disease progression. Lymphopenia or lymphocytopenia is a condition in which the number of lymphocytes in the blood is low. Although T cells can be increased at the onset of COVID-19, these patients tend to have low lymphocyte counts, which is associated with increased COVID-19 severity. Thus, individuals who died of COVID-19 have been shown to have significantly lower lymphocyte levels than survivors. There is evidence that myeloid cells play a role in the pathophysiology of coronavirus infection, either directly as virus targets or indirectly as effectors of cytokine release syndrome. Monocytes are innate hematopoietic cells that maintain vascular homeostasis and provide early responses to pathogens during acute infections. The role of monocytes and macrophages in the resolution of inflammation has also been emphasized as an important component of the response to SARS-CoV-2. Accordingly, it was investigated whether the change observed in blood monocyte levels was an effective parameter in the prognosis process in Covid-19 cases with lymphopenia, considering that monocyte levels could be useful as a guide in the course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Male and female of both genders
* Admitted to the intensive care unit
* Diagnosed with Covid-19 with lymphopenia
* Patients with confirmed COVID-19 diagnosis in polymerase chain reaction (PCR) tests performed on nasopharyngeal swab samples

Exclusion Criteria:

* Those with a negative PCR test
* Aged 18 and under

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted among patients admitted to the intensive care unit of a tertiary hospital.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
prognostic course, rate of mortality | through study completion, an average of 5 month
  The parameters examined will be survival and exitus status, age, weight in kilograms, height in centimeters, weight and height will be combined to report BMI in kg/m^2, gender, presence of additional disease, ferritin, D-dimer, C-reactive protein, lactate dehydrogenase, procalcitonin, fibrinogen, hemoglobin, leukocyte, platelet, neutrophil, eosinophil, basophil, monocyte, lymphocyte levels measured during admission to the intensive care unit. Lymphocyte-monocyte ratio, neutrophil-lymphocyte ratio and platelet-lymphocyte ratio will be obtained from the detected data. The existing O2 requirement at admission to the intensive care unit was recorded retrospectively as fractional inspired oxygen (FiO2) value, the source of oxygen support and the existing Covid-19 treatment. The hemodialysis, vasopressor and intubation requirement that developed during the hospitalization and the exitus status during hospitalization were evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)